CLINICAL TRIAL: NCT04382105
Title: Association Between Salivary IL-6 and Extent of Periodontitis
Brief Title: Evaluation of Saliva IL-6 Levels and Periodontitis
Status: Completed | Type: Observational
Sponsor: University of Messina (Other)
Responsible Party: Principal Investigator, Gaetano Isola, DDS, PhD, Researcher, University of Messina
Other Study IDs: 11-1818
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: observation of salivary IL-6 levels
  Interventions: Other: Observation of salivary IL-6 levels
- Periodontitis: observation of salivary IL-6 levels
  Interventions: Other: Observation of salivary IL-6 levels

INTERVENTIONS:
Other: Observation of salivary IL-6 levels — Observation of salivary IL-6 levels and correlation of salivary IL-6 levels with periodontal disease

SUMMARY:
The aim of this study was to analyze the association between salivary IL-6 levels in patients with periodontitis. Furthermore, the objective was to determine if the periodontitis influenced salivary IL-6 levels

DETAILED DESCRIPTION:
Forty-nine patients with periodontitis and 47 healthy subjects (HS) were enrolled in the present study. Enrolled patients were examined and characterized for clinical and blood samples analysis, and salivary IL-6 levels. The Spearman Correlation Test and Jonckheere-Terpstra Test were applied in order to assess the interdependence between salivary IL-6 levels and clinical periodontal parameters.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least 16 teeth
* CP with a minimum of 40% of sites with a clinical attachment level (CAL)

  ≥2mm and probing depth (PD) ≥4mm;
* Presence of at least ≥2 mm of crestal alveolar bone loss verified on digital periapical radiographs
* Presence of ≥40% sites with bleeding on probing (BOP)

Exclusion Criteria:

* Intake of contraceptives
* Intake of immunosuppressive or anti-inflammatory drugs throughout the last three months prior to the study
* Status of pregnancy or lactation
* Previous history of excessive drinking
* Allergy to local anaesthetic
* Intake of drugs that may potentially determine gingival hyperplasia such as Hydantoin, Nifedipine, Cyclosporin A or similar drugs.

Ages: 35 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Forty-nine patients with periodontitis and 47 healthy subjects (HS) were enrolled in the present study. Enrolled patients were examined and characterized for clinical and blood samples analysis, and salivary P.Gingivalis antibodies were expressed and evaluated enzyme-linked immunosorbent assay (ELISA) units (EU).
Sampling Method: Non-Probability Sample
Enrollment: 287 (Actual)
Dates: Start 2015-11-08 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-09-25 (Actual)

PRIMARY OUTCOMES:
Clinical Attachment Level | 1-year
  evaluation of changes in clinical attachment level

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Matarese, Study Chair — University of Messina
Locations (1):
- University of Messina, Messina, Italy

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: 1-year
Access Criteria: Official website